CLINICAL TRIAL: NCT00037089
Title: A Phase II Study of Paclitaxel, UFT, and Leucovorin in Patients With Metastatic Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Edelman, Martin, M.D. (Individual)
Collaborators: Bristol-Myers Squibb (Industry)
Purpose: Treatment
Other Study IDs: BMS-200604; UMCC 0110g
Record Dates: First submitted 2002-05-14; First posted 2002-05-15 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-01

CONDITIONS: Esophageal Neoplasm
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Tegafur; Uracil

INTERVENTIONS:
Drug: UFT (Tegafur/Uracil)

SUMMARY:
This study is for patients with esophageal cancer that has spread to other areas. The purpose of this study is to:

1. Determine how well a combination of taxol, UFT, and leucovorin work in these patients,
2. Determine the survival of patients with metastatic esophageal carcinoma treated with this combination of drugs.
3. Identify the side effects of this drug combination.

ELIGIBILITY:
INCLUSION

* Histologic proof of esophageal cancer
* No more than one prior non-taxane chemotherapy regimen for either treatment of localized disease or metastatic disease AND they may not have received a regimen containing low dose continuous infusion of 5-FU (i.e. >5 days of infusion/cycle), capecitabine or UFT
* No prior therapy with UFT+/-leucovorin, a taxane, capecitabine, low dose continuous infusion of 5-FU or ethynyl uracil.
* Radiographic or physical examination documentation of metastatic disease
* No major surgery within the 2 weeks preceding the start of treatment and fully recovered from any complications of surgery
* No radiation within 2 weeks of beginning chemotherapy.
* No chemotherapy within 4 weeks of beginning treatment.
* Patients must wait at least 6 weeks after receiving BCNU or Mitomycin-C.
* Minimum life expectancy of 3 months
* Informed consent given
* Laboratory values within limits set by study.

EXCLUSION

* More than one prior chemotherapy regimen for metastatic disease
* Current serious medical or psychiatric illness that would prevent informed consent or intensive treatment
* >grade 1 peripheral sensory or motor neuropathy
* Pregnant
* Patient is taking the drug Sorivudine

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Cancer Center, Baltimore, Maryland, United States